CLINICAL TRIAL: NCT05495087
Title: Intermittent Hypoxia Training: A Novel Therapy for Mild Cognitive Impairment
Brief Title: IHT for Mild Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of North Texas Health Science Center (Other)
Collaborators: University of Texas Southwestern Medical Center (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Xiangrong Shi, Associate Professor, University of North Texas Health Science Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01AG076675 (NIH); R01AG076675 (NIH)
Record Dates: First submitted 2022-07-13; First posted 2022-08-10 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Mild Cognitive Impairment; Memory Impairment
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders

STUDY DESIGN:
Intervention Model Description: IHT vs Sham-IHT Control
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IHT Treatment (Experimental): Exposures to hypoxic air (10% O2) up to 5 min intermittent with up to 5 min recovery (breathing room air) per session, 3 sessions/week, up to 12 weeks.
  Interventions: Device: IHT Treatment
- Sham-IHT control (Placebo Comparator): Exposures to normoxic air (21% O2) up to 5 min intermittent with up to 5 min recovery (breathing room air) per session, 3 sessions/week, up to 12 weeks.
  Interventions: Other: Sham-IHT Control

INTERVENTIONS:
Device: IHT Treatment — IHT Treatment: IH exposure to 10% O2 for up to 5 min, interspersed with breathing room air recovery for up to 5 min, with up to 8 cycles/session, 3 sessions/week, for up to 12 weeks.
  Arms: IHT Treatment
Other: Sham-IHT Control — Sham-IHT Control: Exposure to 21% O2 for up to 5 min, interspersed with breathing room air recovery for up to 5 min, with up to 8 cycles/session, 3 sessions/week, for up to 12 weeks.
  Arms: Sham-IHT control

SUMMARY:
This phase I clinical trial will examine the safety and efficacy of intermittent hypoxia training (IHT) for up to 12 weeks to treat subjects with mild cognitive impairment (MCI).

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women ages 55 to 79 years old who have been diagnosed with MCI.
* Must be willing to be assigned to either group: treatment or sham-treatment control.
* Able to pay multiple visits to the lab for the proposed assessments.
* Able to breathe moderately hypoxic air via an air-cushioned, disposable facemask.
* To have controlled stabilized chronic conditions of at least 6 months duration, such as hypertension, coronary artery disease, diabetes or metabolic disease, chronic bronchitis, degenerative osteoporosis or arthritis and/or other aging-related chronic conditions.
* Must be depression-free at the time of enrollment.
* Must have arterial oxygen saturation at or above 95% and cerebral tissue oxygenation at or above 50% at rest.
* Woman subject must be post-menopausal.

Exclusion Criteria:

* Unwilling to sign a written consent to participate in this double-blinded placebo-controlled phase I trial.
* Diagnosed with AD-dementia or have impaired independent daily functioning; with MMSE <20 and/or CDR ≥1.
* Unable to visit the lab independently.
* Claustrophobic to facemask and hyper-reactive to hypoxia exposure.
* Expecting any major surgery or transplant.
* Have un-controlled chronic conditions including systolic-diastolic pressures over 150/90 mmHg with medications, diabetes, chronic renal failure (based on the medical history questionnaire), obstructive sleep apnea (based on the medical history), recurrent chest pain, seizures or epilepsies, moderate to severe carotid stenosis or calcification, brain aneurysm, uncontrolled allergic rhinitis, pulmonary fibrosis, emphysema, cancer, infectious disease, atrial fibrillation, regular pre-mature ventricular contractions, myocardial ischemia or infarct, 2nd or 3rd degree atrio-ventricular blockade.
* Have severe head injury or traumatic brain injury, stroke (hemorrhagic and/or ischemic).
* Have currently diagnosed depression.
* Currently have COVID-19.
* Have any metallic implants or who are claustrophobic.
* Currently participating in any interventional study and/or have been previously exposed to hypoxia, such as residing more than two months at altitudes above 5000 ft. within the past 3 years or previously participated in a hypoxia training study.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall Cognitive Function | Change from baseline 5-week, 8-week, and up to 12-week intervention
  Change in scores or points (from 0 to 30) in Mini-mental State Examination. Higher scores indicate better testing performance or function.
Attention and Short-term Memory | Change from baseline 5-week, 8-week, and up to 12-week intervention
  Change in scores or points in California-Verbal Learning Test - 2nd edition. Immediate Free-Recall (FR), short-delay FR and long-delay FR for words. More FR words indicate better testing performance and function.
Cognitive Function | Change from baseline 5-week, 8-week, and up to 12-week intervention
  Change in scores or points in Digit-Span test. Two different sets of Forward (from 3 to 9 digits) and Backward (from 2 to 8 digits) Digit-Span recalls test attention and short-term memory. More correct recalls indicate better testing performance and function.
Visual Orientation and Executive Function | Change from baseline 5-week, 8-week, and after up to 12-week intervention
  Change in time to complete Trail-making tests. Less time (in sec) to complete the tests indicates better performance and function.

SECONDARY OUTCOMES:
Neurotoxic Protein | before vs after up to 12-week intervention
  Blood beta-amyloid assessed by enzyme-linked immunosorbent assay. Decreased concentrations indicate a better outcome.
Neuroprotective Protein | before vs after up to 12-week intervention
  Blood erythropoietin assessed by enzyme-linked immunosorbent assay. Increased concentrations indicate a better outcome.
Cerebral Vascular Function | before vs after up to 12-week intervention
  Blood volume flow of carotid artery assessed by ultrasonography. Improved volume flow and vascular compliance in carotid arteries indicate a better outcome.
Brain Morphology | before vs after up to 12-week intervention
  Thickness of cortical gray matter assessed by brain MRI. Increased cerebral cortical gray matter indicates a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Texas Health Science Center, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The summary results information of the trial will be shared, which will include participants' demographic and baseline characteristics, intermittent hypoxia training outcomes (including biosamples data) and statistical analyses, adverse events, and administrative information. All of the submitted results will be de-identified; no participant ID or identifiable information will be included in the shared results information.
Supporting Information: SAP, CSR
Time Frame: 9 months after publication of major data for 3 years
Access Criteria: Sharing the data by creating a record of the study in the Global Alzheimer's Association interactive Network (GAAIN.org).